CLINICAL TRIAL: NCT04360863
Title: The Impact of Coronavirus Disease (COVID-19) Pandemic on the Smoking Behaviour of Young Smokers and the Youth Quitline Service in Hong Kong: A Survey Study
Brief Title: The Impact of COVID-19 Pandemic on the Smoking Behaviour of Young Smokers and the Youth Quitline Service in Hong Kong
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Other Study IDs: NCT02758028_1
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Smoking Cessation
Keywords: Youth smokers; COVID-19; smoking behaviors
MeSH Terms: conditions — Smoking Cessation; COVID-19; Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Youth smokers: Participants of Youth Quitline
  Interventions: Other: Telephone survey

INTERVENTIONS:
Other: Telephone survey — Participants will be asked to respond to a survey regarding their knowledge about the relationship between smoking and COVID-19, their smoking behaviors and readiness to quit during the pandemic.

SUMMARY:
The aims of the present study are:

1. To explore the impact of COVID-19 pandemic on the smoking behavior of youth smokers
2. To explore the impact of COVID-19 pandemic on the Youth Quitline service in Hong Kong

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) pandemic has spread rapidly across the globe. According to World Health Organization (WHO), due to the harmful effects on the lungs and the possible viral transmission from fingers to mouth during smoking, tobacco use is considered a major risk factor for developing COVID-19. Both tobacco use and COVID-19 can cause damage to the cardiovascular and respiratory systems. Smokers infected with COVID-19 are at higher risk of developing severe COVID-19 symptoms or death than non-smokers.

The Hong Kong SAR (HKSAR) government has announced different regulations to combat the spread of COVID-19 since late January 2020, which significantly affect the working patterns and everyday lives of people. It remains unknown how smoking habits and smoking cessation services are being affected during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong resident aged 25 or below
* Able to communicate in Chinese (Cantonese)
* Smoked in the past 30 days

Exclusion Criteria:

* Have difficulty to communicate via telephone

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Youth smokers
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Smoking behaviors | Baseline
  Change in smoking behaviors of youth smokers during the pandemic
Knowledge | Baseline
  Knowledge regarding the relationship between COVID-19 and smoking
Readiness to quit | Baseline
  Change in motivation to quit during the pandemic

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project is completed and the results of the project has been published.
Access Criteria: Request could be sent to Principal Investigator (william3@hku.hk)